CLINICAL TRIAL: NCT01856543
Title: Mometasone Furoate 0.1% Versus Eucerin on Moderate to Severe Skin Toxicities in Breast Cancer Patients Receiving Postmastectomy Radiation:A Randomized Trial, Double Blind Trial
Brief Title: Mometasone Furoate 0.1% Versus Eucerin on Moderate to Severe Skin Toxicities in Breast Cancer Patients Receiving Postmastectomy Radiation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-069
Record Dates: First submitted 2013-05-15; First posted 2013-05-17 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2018-08

CONDITIONS: Invasive Breast Cancer
Keywords: Breast cancer; Status post mastectomy; plan to receive PMRT; Topical; steroid cream; emollient skin care; Eucerin; Mometasone Furoate 0.1%
MeSH Terms: conditions — Breast Neoplasms | interventions — eucerin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Eucerin (Placebo Comparator): Patient education regarding amount to be applied (amount depending on body habitus) and area of treatment field will be reinforced by the R.N. prior to the first radiation treatment. Part of patient education may involve application of the cream. Patients will be instructed to apply cream to the upper outer quadrant, upper inner quadrant, lower outer quadrant, and lower inner quadrant, as well as irradiated nodal fields. They will be instructed to apply cream in a thin, uniform layer twice a day, in the morning and evening, and not within the immediate 4 hours prior to radiation treatment. Patients will be informed that application immediately following radiation treatment is acceptable for those scheduled to receive morning treatments. Patients will be provided diaries to record the date and time they applied the study cream. Pts should return the completed diaries on their weekly status checks and at the 2 weeks +/- 2 business days following the completion of RT.
  Interventions: Other: Eucerin
- Mometasone Furoate 0.1% (Experimental): Patient education regarding amount to be applied (amount depending on body habitus) and area of treatment field will be reinforced by the R.N. prior to the first radiation treatment. Part of patient education may involve application of the cream. Patients will be instructed to apply cream to the upper outer quadrant, upper inner quadrant, lower outer quadrant, and lower inner quadrant, as well as irradiated nodal fields. They will be instructed to apply cream in a thin, uniform layer twice a day, in the morning and evening, and not within the immediate 4 hours prior to radiation treatment. Patients will be informed that application immediately following radiation treatment is acceptable for those scheduled to receive morning treatments. Patients will be provided diaries to record the date and time they applied the study cream. Patients should return the completed diaries on their weekly status checks and at the 2 weeks +/- 2 business days following the completion of RT.
  Interventions: Other: Mometasone Furoate 0.1%

INTERVENTIONS:
Other: Eucerin
  Arms: Eucerin
Other: Mometasone Furoate 0.1%
  Arms: Mometasone Furoate 0.1%

SUMMARY:
The purpose of this study is to find out if the effect of mometasone furoate is any different from Eucerin in decreasing the severity of redness of the skin during irradiation, preventing the skin from peeling, or reducing the amount of irritation the patient reports during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Stage 1-4 invasive breast cancer that is histologically confirmed at MSKCC
* Status post mastectomy with axillary exploration (sentinel node biopsy and/or axillary lymph node dissection) to receive PMRT
* ECOG Performance Status of 0 or 1

Exclusion Criteria:

* Male
* Patients with clinical evidence of gross disease
* Patients who are pregnant or breastfeeding
* Prior radiation therapy to the ipsilateral chest wall or thorax
* Patients requiring a chest wall boost
* Concurrent chemotherapy (biologic agents are allowed)
* Psychiatric illness that would prevent the patient from giving informed consent
* Inability or unwillingness to comply with skin care instructions and follow-up
* Allergy to either Eucerin or MF
* Residual grade >1 skin toxicity, cellulitis, or incompletely healed wound(s) at intended site of study drug application at the time of the start of RT
* Medical condition such as uncontrolled infection (including HIV), uncontrolled diabetes mellitus, or connective tissue diseases (lupus, systemic sclerosis, or other collagen vascular diseases)
* Treatment with palliative or pre-operative radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Molly Olm-Shipman, RN, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Eucerin: Patient education regarding amount to be applied (amount depending on body habitus) and area of treatment field will be reinforced by the R.N. prior to the first radiation treatment. Part of patient education may involve application of the cream. Patients will be instructed to apply cream to the upper outer quadrant, upper inner quadrant, lower outer quadrant, and lower inner quadrant, as well as irradiated nodal fields. They will be instructed to apply cream in a thin, uniform layer twice a day, in the morning and evening, and not within the immediate 4 hours prior to radiation treatment. Patients will be informed that application immediately following radiation treatment is acceptable for those scheduled to receive morning treatments. Patients will be provided diaries to record the date and time they applied the study cream. Pts should return the completed diaries on their weekly status checks and at the 2 weeks +/- 2 business days following the completion of RT.
  Eucerin
- Mometasone Furoate 0.1%: Patient education regarding amount to be applied (amount depending on body habitus) and area of treatment field will be reinforced by the R.N. prior to the first radiation treatment. Part of patient education may involve application of the cream. Patients will be instructed to apply cream to the upper outer quadrant, upper inner quadrant, lower outer quadrant, and lower inner quadrant, as well as irradiated nodal fields. They will be instructed to apply cream in a thin, uniform layer twice a day, in the morning and evening, and not within the immediate 4 hours prior to radiation treatment. Patients will be informed that application immediately following radiation treatment is acceptable for those scheduled to receive morning treatments.
  Mometasone F
Period: Overall Study
Arm/Group | Eucerin | Mometasone Furoate 0.1%
Started | 73 | 70
Completed | 60 | 64
Not Completed | 13 | 6
Not completed — Treatment discontinued | 6 | 3
Not completed — Withdrawn before start | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eucerin | Mometasone Furoate 0.1% | Total
Number analyzed (Participants) | 73 | 70 | 143
Age, Continuous [Mean (Full Range); unit: years] | 49 [26 to 80] | 48 [26 to 76] | 49 [26 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 70 | 143
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 12 | 25
  White | 49 | 46 | 95
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 5 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 73 | 70 | 143

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Moist Desquamation
Description: Skin toxicity assessments will be done on a weekly basis while the patient is receiving RT, by the RN or physician utilizing CTCAE 4.0 and the weekly status check form, as per current standard practice.
Time Frame: 2 years
Measure: Number; unit: % of participants w/moist desquamation
Arm/Group | Eucerin | Mometasone Furoate 0.1%
Number analyzed (Participants) | 73 | 70
% of participants w/moist desquamation | 66.7 | 43.8

2. Secondary Outcome: Difference From Baseline and 5 Weeks Between Patient-reported Skin Toxicities at Baseline and End of Radiation Treatment
Description: The Skindex-16 assessment tool is designed to capture patient-reported assessments of subjective adverse effects. It consists of a short 16-item assessment completed by the patient, with each item rated on a 7-point Likert scale (0=never bothered to 6=always bothered). Responses to the Skindex-16 are categorized into three subscales: symptom, emotional, and functional. Scores for the emotions, symptoms and functioning scales are also expressed in a linear scale from 0 to 100. Rankings of the questionnaire are then averaged to obtain a score of severity of patient-reported outcomes. This allows providers to gauge which aspects of the participant's experience are most affected by the treatment.
Time Frame: 5 weeks and Baseline
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- Mometasone Furoate 0.1%: Patient education regarding amount to be applied (amount depending on body habitus) and area of treatment field will be reinforced by the R.N. prior to the first radiation treatment. Part of patient education may involve application of the cream. Patients will be instructed to apply cream to the upper outer quadrant, upper inner quadrant, lower outer quadrant, and lower inner quadrant, as well as irradiated nodal fields. They will be instructed to apply cream in a thin, uniform layer twice a day, in the morning and evening, and not within the immediate 4 hours prior to radiation treatment. Patients will be informed that application immediately following radiation treatment is acceptable for those scheduled to receive morning treatments.
Arm/Group | Eucerin | Mometasone Furoate 0.1%
Number analyzed (Participants) | 60 | 64
score on a scale
  Emotions | 8.0 (11.4) | 5.0 (9.1)
  Symptoms | 6.0 (7.2) | 6.0 (6.4)
  Functioning | 2.0 (7.4) | 1.0 (5.3)

3. Secondary Outcome: Difference Between Patient-reported Skin Toxicities at End of Radiation Therapy and 2 Week Follow-up
Description: as for outcome 2
Time Frame: 2 weeks after end of Radiation Therapy
Measure: Median (Standard Deviation); unit: scores on a scale
Arm/Group | Eucerin | Mometasone Furoate 0.1%
Number analyzed (Participants) | 60 | 64
scores on a scale
  Emotions | 15.0 (12.3) | 12.0 (12.8)
  Symptoms | 11.0 (7.4) | 11.0 (6.7)
  Functioning | 6.0 (7.9) | 5.0 (9.1)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Eucerin | Mometasone Furoate 0.1%
All-Cause Mortality (participants affected / at risk) | 5/73 | 6/70
Serious Adverse Events (participants affected / at risk) | 3/73 | 3/70
Other Adverse Events (participants affected / at risk) | 25/73 | 29/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eucerin (N=73) | Mometasone Furoate 0.1% (N=70)
Chest Pain - cardiac (Cardiac disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 1
Skin infection (Infections and infestations) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eucerin (N=73) | Mometasone Furoate 0.1% (N=70)
Lymphocyte count decreased (Investigations) | 13 | 10
White blood cell decreased (Investigations) | 6 | 8
Dermatitis radiation (Injury, poisoning and procedural complications) | 4 | 1
Neutrophil count decreased (Investigations) | 1 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT01856543/Prot_SAP_000.pdf